CLINICAL TRIAL: NCT03093623
Title: The Effect of Physical Activity and Abstain From Smoking on the Regression of Precancerous Lesion.
Brief Title: The Effect of Physical Activity and Abstain From Smoking on the Precancerous Lesion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: TMU-JIRB:201410013
Record Dates: First submitted 2017-03-23; First posted 2017-03-28 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2016-12

CONDITIONS: Cancer Cervix Uterus; Precancerous Lesions; Smoking
Keywords: physical activity; abstain from smoking; human papillomavirus (HPV); cervical intraepithelial neoplasia (CIN)
MeSH Terms: conditions — Smoking; Motor Activity; Uterine Cervical Dysplasia | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity (Experimental): In physical activity experimental group, trained study nurses will interview with patients,give health education,teach how to use and record the Activity meter.Professionals will calculate Metabolic Equivalent of Task(MET) with formula weekly.MET = (intensity level 9 points * time of each exercise (hours) * Number of times per week + moderate level 5 points * time per activity (hours) * number of times per week + low level 3 points * time per activity (hours) * number of times per week),investigators hope patients in the first month MET can reach (3.75-7.49 MET-h/ week), and reach moderate or more than moderate activity (>= 7.5-16.49 MET-h/ week) at the starting of second month for at least one year.
  Interventions: Behavioral: Physical activity
- Non-Physical activity (No Intervention): the non-physical activity group,investigators do not give them any physical interventions

INTERVENTIONS:
Behavioral: Physical activity — In physical activity experimental group, trained study nurses will interview with patients,give health education,teach how to use and record the Activity meter.Professionals will calculate Metabolic Equivalent of Task(MET) with formula weekly.MET = (intensity level 9 points * time of each exercise (hours) * Number of times per week + moderate level 5 points * time per activity (hours) * number of times per week + low level 3 points * time per activity (hours) * number of times per week),investigators hope patients in the first month MET can reach (3.75-7.49 MET-h/ week), and reach moderate or more than moderate activity (>= 7.5-16.49 MET-h/ week) at the starting of second month for at least one year.
  Arms: Physical activity

SUMMARY:
In this proposed project,investigators will estimate the effect of physical activity and abstain from smoking on the regression of precancerous neoplasia.

DETAILED DESCRIPTION:
Cervical cancer is the seventh most common malignancy and the sixth most common cause of cancer-related death in Taiwan. The development of cervical cancer is passed through cervical intraepithelial neoplasia (CIN), including CIN I, CIN II, and CIN III. CIN I is classified as low-grade squamous intraepithelial lesion (LSIL), and about 57% of patients with CIN I are known to regress spontaneously, while patients with CIN II or CIN III is 5% and 15% to progress to invasive cervical cancer, respectively. Both two need active treatment and are classified as high-grade squamous intraepithelial lesion (HSIL). Fortunately, the 5-year survival rate is more than 90% for patients with CINs if they receive clinical management as soon as possible. The immunocompetence plays an important role for prevention of cervical cancer. High-risk human papillomavirus (HR-HPV) infection is demonstrated as one of the vital risk factors of CIN and cervical cancer. Most HPV infection is known to regress spontaneously by cell-mediated immunity, whereas a small fraction persistant HPV infection, which increase the risk of CIN and promote the progression to cervical cancer. Physical activity is reported to increase the cell number and activity of immune cells and promote cell-mediated cytotoxic effect to protect against HPV and cancer cells. Also, it is found that physical activity decrease the risk of breast cancer, hepatocellular carcinoma, colon cancer, and prostate cancer. Regular moderate intensity physical activity is ssociated with a decrease in the death from cancer. Moreover, tobacco smoke is reported to abate human immunocompetence and raise the risk of cervical cancer as well as to enhance the progression of CIN through the inhibition of cell-mediated immunity. Also, the extract of tobacco is demonstrated to enhance the proliferation and viral load of HPV, consequently induce carcinogenesis of cervical intraepithelial cells. Investigators suggest that physical activity could decrease the risk of CIN through promote cell-mediated immunity. Also, physical activity and abstain from smoking could be benefit to the regression of CIN and the decreasing of DNA viral load of HPV. However, the roles of physical activity and abstain from smoking on the regression of CIN and viral load are not fully clarified. Therefore, in this proposed project, investigators will 【1】estimate the effect of physical activity on decreasing the risk of cervical intraepithelial neoplasia. 【2】estimate the effect of physical activity on the regression of cervical intraepithelial neoplasia. 【3】estimate the effect of abstain from smoking on the regression of cervical intraepithelial neoplasia. 【4】estimate the additive effect and synergistic effect of physical activity and abstain from smoking on the regression of cervical intraepithelial neoplasia. 【5】estimate the effect of physical activity on the decreasing of DNA viral load of human papillomavirus. 【6】estimate the effect of abstain from smoking on the decreasing of DNA viral load of human papillomavirus. 【7】estimate the additive effect and synergistic effect of physical activity and abstain from smoking on the decreasing of DNA viral load of human papillomavirus

ELIGIBILITY:
Inclusion Criteria:

* Patients with precancerous neoplasia
* between 20 to 70 years

Exclusion Criteria:

* Patients with server heart disease or other cancer.

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The effect of physical activity and abstain from smoking on the regression of precancerous | 2 years
  To estimate the effect of moderate physical activity and abstain from smoking can strengthen the innate immune system,adaptive human immune system and can help regression of Cervical intraepithelial neoplasia among patients with cervical cancer.
  Using a composite outcome measure consisting of questionnaire,blood counts,plasma and DNA.
  blood counts :white blood cells,hemoglobin,red blood cells,platelets,Neutrophil,Lymphocyte,Monocyte,Eosinophil,Basophil,CD-4,CD-8,NK-cell,B-cell.
  plasma:lL-1,IL-2,IL-4,IL-5,IL,6,LI-8,IL-10,IL-13,TNF-r

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Ting Tsai, Phd, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ye F, Chen S, Liu W. Effects of electro-acupuncture on immune function after chemotherapy in 28 cases. J Tradit Chin Med. 2002 Mar;22(1):21-3. PMID 11977512
- [Result] Wen CP, Wai JP, Tsai MK, Yang YC, Cheng TY, Lee MC, Chan HT, Tsao CK, Tsai SP, Wu X. Minimum amount of physical activity for reduced mortality and extended life expectancy: a prospective cohort study. Lancet. 2011 Oct 1;378(9798):1244-53. doi: 10.1016/S0140-6736(11)60749-6. Epub 2011 Aug 16. PMID 21846575
- [Result] http://www.health.gov/paguidelines/committeereport.aspx.
- [Result] Goh J, Kirk EA, Lee SX, Ladiges WC. Exercise, physical activity and breast cancer: the role of tumor-associated macrophages. Exerc Immunol Rev. 2012;18:158-76. PMID 22876727
- [Result] Mason C, Alfano CM, Smith AW, Wang CY, Neuhouser ML, Duggan C, Bernstein L, Baumgartner KB, Baumgartner RN, Ballard-Barbash R, McTiernan A. Long-term physical activity trends in breast cancer survivors. Cancer Epidemiol Biomarkers Prev. 2013 Jun;22(6):1153-61. doi: 10.1158/1055-9965.EPI-13-0141. Epub 2013 Apr 10. PMID 23576689
- [Result] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Result] Singh AA, Jones LW, Antonelli JA, Gerber L, Calloway EE, Shuler KH, Freedland SJ, Grant DJ, Hoyo C, Banez LL. Association between exercise and primary incidence of prostate cancer: does race matter? Cancer. 2013 Apr 1;119(7):1338-43. doi: 10.1002/cncr.27791. Epub 2013 Feb 11. PMID 23401030
- [Result] Santoso JT, Crigger M, English E, Wan J, Likes W. Smoking cessation counseling in women with genital intraepithelial neoplasia. Gynecol Oncol. 2012 Jun;125(3):716-9. doi: 10.1016/j.ygyno.2012.02.018. Epub 2012 Feb 21. PMID 22366589
- [Result] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Result] Behrens G, Matthews CE, Moore SC, Freedman ND, McGlynn KA, Everhart JE, Hollenbeck AR, Leitzmann MF. The association between frequency of vigorous physical activity and hepatobiliary cancers in the NIH-AARP Diet and Health Study. Eur J Epidemiol. 2013 Jan;28(1):55-66. doi: 10.1007/s10654-013-9767-1. Epub 2013 Jan 26. PMID 23354983
- [Result] Wu Y, Zhang D, Kang S. Physical activity and risk of breast cancer: a meta-analysis of prospective studies. Breast Cancer Res Treat. 2013 Feb;137(3):869-82. doi: 10.1007/s10549-012-2396-7. Epub 2012 Dec 30. PMID 23274845
- [Result] Beesley VL, Eakin EG, Janda M, Battistutta D. Gynecological cancer survivors' health behaviors and their associations with quality of life. Cancer Causes Control. 2008 Sep;19(7):775-82. doi: 10.1007/s10552-008-9140-y. Epub 2008 Mar 6. PMID 18322812
- [Result] Buffart LM, Galvao DA, Chinapaw MJ, Brug J, Taaffe DR, Spry N, Joseph D, Newton RU. Mediators of the resistance and aerobic exercise intervention effect on physical and general health in men undergoing androgen deprivation therapy for prostate cancer. Cancer. 2014 Jan 15;120(2):294-301. doi: 10.1002/cncr.28396. Epub 2013 Oct 7. PMID 24122296
- [Result] Gho SA, Steele JR, Jones SC, Munro BJ. Self-reported side effects of breast cancer treatment: a cross-sectional study of incidence, associations, and the influence of exercise. Cancer Causes Control. 2013 Mar;24(3):517-28. doi: 10.1007/s10552-012-0142-4. Epub 2013 Jan 8. PMID 23296457
- [Result] Rausch SM, Millay S, Scott C, Pruthi S, Clark MM, Patten C, Stan D, Sellers T, Vachon C. Health behaviors among cancer survivors receiving screening mammography. Am J Clin Oncol. 2012 Feb;35(1):22-31. doi: 10.1097/COC.0b013e318200598e. PMID 21293247
- [Result] Inamine M, Nagai Y, Mitsuhashi A, Nagase S, Yaegashi N, Yoshikawa H, Aoki Y. Cigarette smoke stimulates VEGF-C expression in cervical intraepithelial neoplasia (CIN) 1 and 2 lesions. Int J Clin Oncol. 2012 Oct;17(5):498-504. doi: 10.1007/s10147-011-0322-3. Epub 2011 Sep 27. PMID 21947598
- [Result] Matsumoto K, Oki A, Furuta R, Maeda H, Yasugi T, Takatsuka N, Hirai Y, Mitsuhashi A, Fujii T, Iwasaka T, Yaegashi N, Watanabe Y, Nagai Y, Kitagawa T, Yoshikawa H; Japan HPV And Cervical Cancer (JHACC) Study Group. Tobacco smoking and regression of low-grade cervical abnormalities. Cancer Sci. 2010 Sep;101(9):2065-73. doi: 10.1111/j.1349-7006.2010.01642.x. PMID 20626752
- [Result] Szarewski A, Jarvis MJ, Sasieni P, Anderson M, Edwards R, Steele SJ, Guillebaud J, Cuzick J. Effect of smoking cessation on cervical lesion size. Lancet. 1996 Apr 6;347(9006):941-3. doi: 10.1016/s0140-6736(96)91417-8. PMID 8598759
- [Result] Karst M, Schneidewind D, Scheinichen D, Juettner B, Bernateck M, Molsberger A, Parlesak A, Passie T, Hoy L, Fink M. Acupuncture induces a pro-inflammatory immune response intensified by a conditioning-expectation effect. Forsch Komplementmed. 2010 Mar;17(1):21-7. doi: 10.1159/000264657. Epub 2010 Mar 4. PMID 20215759
- [Result] Pavao TS, Vianna P, Pillat MM, Machado AB, Bauer ME. Acupuncture is effective to attenuate stress and stimulate lymphocyte proliferation in the elderly. Neurosci Lett. 2010 Oct 22;484(1):47-50. doi: 10.1016/j.neulet.2010.08.016. Epub 2010 Aug 13. PMID 20709154
- [Result] Kou W, Bell JD, Gareus I, Pacheco-Lopez G, Goebel MU, Spahn G, Stratmann M, Janssen OE, Schedlowski M, Dobos GJ. Repeated acupuncture treatment affects leukocyte circulation in healthy young male subjects: a randomized single-blind two-period crossover study. Brain Behav Immun. 2005 Jul;19(4):318-24. doi: 10.1016/j.bbi.2004.10.001. Epub 2004 Nov 25. PMID 15944071
- [Result] Lin GJ, Fat u Camar a. [Randomized and controlled observation on acupuncture and moxibustion combined with western medicine for treatment of malaria of children in Africa]. Zhongguo Zhen Jiu. 2007 Nov;27(11):859-61. Chinese. PMID 18085153
- [Result] Ishikawa S, Murai M, Sato T, Sunagawa M, Tokita E, Aung SK, Asano K, Hisamitsu T. Promotion of blood fluidity by inhibition of platelet adhesion using electroacupuncture stimulation. J Acupunct Meridian Stud. 2011 Mar;4(1):44-53. doi: 10.1016/S2005-2901(11)60006-X. PMID 21440879
- [Result] Ishikawa S, Suga H, Fukushima M, Yoshida A, Yoshida Y, Sunagawa M, Hisamitsu T. Blood fluidity enhancement by electrical acupuncture stimulation is related to an adrenergic mechanism. J Acupunct Meridian Stud. 2012 Feb;5(1):21-8. doi: 10.1016/j.jams.2011.11.003. Epub 2011 Dec 17. PMID 22309904
- [Result] http://www.cdc.gov/physicalactivity.
- [Result] Department of Health: Republic of China: ''Health Promotion Administration, Ministry of Health and Welfare'' Department of Health. Taipei 2013
- [Result] Steele JC, Mann CH, Rookes S, Rollason T, Murphy D, Freeth MG, Gallimore PH, Roberts S. T-cell responses to human papillomavirus type 16 among women with different grades of cervical neoplasia. Br J Cancer. 2005 Jul 25;93(2):248-59. doi: 10.1038/sj.bjc.6602679. PMID 15986031
- [Result] Stanley MA. Immune responses to human papilloma viruses. Indian J Med Res. 2009 Sep;130(3):266-76. PMID 19901436
- [Result] Sasagawa T, Takagi H, Makinoda S. Immune responses against human papillomavirus (HPV) infection and evasion of host defense in cervical cancer. J Infect Chemother. 2012 Dec;18(6):807-15. doi: 10.1007/s10156-012-0485-5. Epub 2012 Nov 3. PMID 23117294
- [Result] Huang CY, Chen JJ, Shen KY, Chang LS, Yeh YC, Chen IH, Chong P, Liu SJ, Leng CH. Recombinant lipidated HPV E7 induces a Th-1-biased immune response and protective immunity against cervical cancer in a mouse model. PLoS One. 2012;7(7):e40970. doi: 10.1371/journal.pone.0040970. Epub 2012 Jul 18. PMID 22815882
- [Result] Feng Q, Wei H, Morihara J, Stern J, Yu M, Kiviat N, Hellstrom I, Hellstrom KE. Th2 type inflammation promotes the gradual progression of HPV-infected cervical cells to cervical carcinoma. Gynecol Oncol. 2012 Nov;127(2):412-9. doi: 10.1016/j.ygyno.2012.07.098. Epub 2012 Jul 22. PMID 22828962
- [Result] Welters MJ, van der Logt P, van den Eeden SJ, Kwappenberg KM, Drijfhout JW, Fleuren GJ, Kenter GG, Melief CJ, van der Burg SH, Offringa R. Detection of human papillomavirus type 18 E6 and E7-specific CD4+ T-helper 1 immunity in relation to health versus disease. Int J Cancer. 2006 Feb 15;118(4):950-6. doi: 10.1002/ijc.21459. PMID 16152582
- [Result] Peghini BC, Abdalla DR, Barcelos AC, Teodoro Ld, Murta EF, Michelin MA. Local cytokine profiles of patients with cervical intraepithelial and invasive neoplasia. Hum Immunol. 2012 Sep;73(9):920-6. doi: 10.1016/j.humimm.2012.06.003. Epub 2012 Jun 28. PMID 22749886
- [Result] Tsai HT, Wu CH, Lai HL, Li RN, Tung YC, Chuang HY, Wu TN, Lin LJ, Ho CK, Liu HW, Wu MT. Association between quantitative high-risk human papillomavirus DNA load and cervical intraepithelial neoplasm risk. Cancer Epidemiol Biomarkers Prev. 2005 Nov;14(11 Pt 1):2544-9. doi: 10.1158/1055-9965.EPI-05-0240. PMID 16284376
- [Result] Garcia-Iglesias T, Del Toro-Arreola A, Albarran-Somoza B, Del Toro-Arreola S, Sanchez-Hernandez PE, Ramirez-Duenas MG, Balderas-Pena LM, Bravo-Cuellar A, Ortiz-Lazareno PC, Daneri-Navarro A. Low NKp30, NKp46 and NKG2D expression and reduced cytotoxic activity on NK cells in cervical cancer and precursor lesions. BMC Cancer. 2009 Jun 16;9:186. doi: 10.1186/1471-2407-9-186. PMID 19531227
- [Result] Balkwill F, Mantovani A. Inflammation and cancer: back to Virchow? Lancet. 2001 Feb 17;357(9255):539-45. doi: 10.1016/S0140-6736(00)04046-0. PMID 11229684
- [Result] Azar KK, Tani M, Yasuda H, Sakai A, Inoue M, Sasagawa T. Increased secretion patterns of interleukin-10 and tumor necrosis factor-alpha in cervical squamous intraepithelial lesions. Hum Pathol. 2004 Nov;35(11):1376-84. doi: 10.1016/j.humpath.2004.08.012. PMID 15668895
- [Result] Bermudez-Morales VH, Gutierrez LX, Alcocer-Gonzalez JM, Burguete A, Madrid-Marina V. Correlation between IL-10 gene expression and HPV infection in cervical cancer: a mechanism for immune response escape. Cancer Invest. 2008 Dec;26(10):1037-43. doi: 10.1080/07357900802112693. PMID 18798072
- [Result] Bolpetti A, Silva JS, Villa LL, Lepique AP. Interleukin-10 production by tumor infiltrating macrophages plays a role in Human Papillomavirus 16 tumor growth. BMC Immunol. 2010 Jun 7;11:27. doi: 10.1186/1471-2172-11-27. PMID 20525400
- [Result] Maddocks M, Jones LW, Wilcock A. Immunological and hormonal effects of exercise: implications for cancer cachexia. Curr Opin Support Palliat Care. 2013 Dec;7(4):376-82. doi: 10.1097/SPC.0000000000000010. PMID 24157716
- [Result] Bigley AB, Spielmann G, LaVoy EC, Simpson RJ. Can exercise-related improvements in immunity influence cancer prevention and prognosis in the elderly? Maturitas. 2013 Sep;76(1):51-6. doi: 10.1016/j.maturitas.2013.06.010. Epub 2013 Jul 17. PMID 23870832
- [Result] Kruijsen-Jaarsma M, Revesz D, Bierings MB, Buffart LM, Takken T. Effects of exercise on immune function in patients with cancer: a systematic review. Exerc Immunol Rev. 2013;19:120-43. PMID 23977724
- [Result] Shimizu K, Suzuki N, Imai T, Aizawa K, Nanba H, Hanaoka Y, Kuno S, Mesaki N, Kono I, Akama T. Monocyte and T-cell responses to exercise training in elderly subjects. J Strength Cond Res. 2011 Sep;25(9):2565-72. doi: 10.1519/JSC.0b013e3181fc5e67. PMID 21685807
- [Result] Rogers CJ, Colbert LH, Greiner JW, Perkins SN, Hursting SD. Physical activity and cancer prevention : pathways and targets for intervention. Sports Med. 2008;38(4):271-96. doi: 10.2165/00007256-200838040-00002. PMID 18348589
- [Result] Spielmann G, McFarlin BK, O'Connor DP, Smith PJ, Pircher H, Simpson RJ. Aerobic fitness is associated with lower proportions of senescent blood T-cells in man. Brain Behav Immun. 2011 Nov;25(8):1521-9. doi: 10.1016/j.bbi.2011.07.226. Epub 2011 Jul 19. PMID 21784146
- [Result] Hayes SC, Rowbottom D, Davies PS, Parker TW, Bashford J. Immunological changes after cancer treatment and participation in an exercise program. Med Sci Sports Exerc. 2003 Jan;35(1):2-9. doi: 10.1097/00005768-200301000-00002. PMID 12544628
- [Result] Kim SD, Kim HS. A series of bed exercises to improve lymphocyte count in allogeneic bone marrow transplantation patients. Eur J Cancer Care (Engl). 2006 Dec;15(5):453-7. doi: 10.1111/j.1365-2354.2006.00668.x. PMID 17177902
- [Result] IARC Monographs programme on the evaluation of the carcinogenic risk of chemicals to humans. Preamble. IARC Monogr Eval Carcinog Risk Chem Hum. 1986;39:13-32. No abstract available. PMID 3465680
- [Result] Jacobsen PB, Phillips KM, Jim HS, Small BJ, Faul LA, Meade CD, Thompson L, Williams CC Jr, Loftus LS, Fishman M, Wilson RW. Effects of self-directed stress management training and home-based exercise on quality of life in cancer patients receiving chemotherapy: a randomized controlled trial. Psychooncology. 2013 Jun;22(6):1229-35. doi: 10.1002/pon.3122. Epub 2012 Jun 20. PMID 22715124
- [Result] Prokopczyk B, Cox JE, Hoffmann D, Waggoner SE. Identification of tobacco-specific carcinogen in the cervical mucus of smokers and nonsmokers. J Natl Cancer Inst. 1997 Jun 18;89(12):868-73. doi: 10.1093/jnci/89.12.868. PMID 9196253
- [Result] Sizemore N, Mukhtar H, Couch LH, Howard PC, Rorke EA. Differential response of normal and HPV immortalized ectocervical epithelial cells to B[a]P. Carcinogenesis. 1995 Oct;16(10):2413-8. doi: 10.1093/carcin/16.10.2413. PMID 7586144
- [Result] Anisimov VN, Zabezhinski MA, Popovich IG, Zaripova EA, Musatov SA, Andre V, Vigreux C, Godard T, Sichel F. Inhibitory effect of melatonin on 7, 12-dimethylbenz[a]anthracene-induced carcinogenesis of the uterine cervix and vagina in mice and mutagenesis in vitro. Cancer Lett. 2000 Aug 11;156(2):199-205. doi: 10.1016/s0304-3835(00)00463-8. PMID 10880770
- [Result] Kaufman DW, Palmer JR, Rosenberg L, Stolley P, Warshauer E, Shapiro S. Tar content of cigarettes in relation to lung cancer. Am J Epidemiol. 1989 Apr;129(4):703-11. doi: 10.1093/oxfordjournals.aje.a115185. PMID 2923118
- [Result] Clarke EA, Morgan RW, Newman AM. Smoking as a risk factor in cancer of the cervix: additional evidence from a case-control study. Am J Epidemiol. 1982 Jan;115(1):59-66. doi: 10.1093/oxfordjournals.aje.a113279. PMID 7055130
- [Result] Coker AL, Rosenberg AJ, McCann MF, Hulka BS. Active and passive cigarette smoke exposure and cervical intraepithelial neoplasia. Cancer Epidemiol Biomarkers Prev. 1992 Jul-Aug;1(5):349-56. PMID 1305466
- [Result] Gram IT, Austin H, Stalsberg H. Cigarette smoking and the incidence of cervical intraepithelial neoplasia, grade III, and cancer of the cervix uteri. Am J Epidemiol. 1992 Feb 15;135(4):341-6. doi: 10.1093/oxfordjournals.aje.a116295. PMID 1550088
- [Result] Wu MT, Lee LH, Ho CK, Liu CL, Wu TN, Wu SC, Lin LY, Cheng BH, Yang CY. Lifetime exposure to environmental tobacco smoke and cervical intraepithelial neoplasms among nonsmoking Taiwanese women. Arch Environ Health. 2003 Jun;58(6):353-9. PMID 14992310
- [Result] Tsai HT, Tsai YM, Yang SF, Wu KY, Chuang HY, Wu TN, Ho CK, Lin CC, Kuo YS, Wu MT. Lifetime cigarette smoke and second-hand smoke and cervical intraepithelial neoplasm--a community-based case-control study. Gynecol Oncol. 2007 Apr;105(1):181-8. doi: 10.1016/j.ygyno.2006.11.012. Epub 2007 Jan 3. PMID 17204311
- [Result] Girianelli VR, Azevedo E Silva G, Thuler LC. Factors associated with the risk of progression to precursor lesions or cervical cancer in women with negative cytologic findings. Int J Gynaecol Obstet. 2009 Dec;107(3):228-31. doi: 10.1016/j.ijgo.2009.07.036. Epub 2009 Aug 28. PMID 19716561
- [Result] Poppe WA, Ide PS, Drijkoningen MP, Lauweryns JM, Van Assche FA. Tobacco smoking impairs the local immunosurveillance in the uterine cervix. An immunohistochemical study. Gynecol Obstet Invest. 1995;39(1):34-8. doi: 10.1159/000292372. PMID 7890250
- [Result] Castellsague X, Munoz N. Chapter 3: Cofactors in human papillomavirus carcinogenesis--role of parity, oral contraceptives, and tobacco smoking. J Natl Cancer Inst Monogr. 2003;(31):20-8. PMID 12807941
- [Result] Montoya L. Managing hematologic toxicities in the oncology patient. J Infus Nurs. 2007 May-Jun;30(3):168-72. doi: 10.1097/01.NAN.0000270676.59180.c3. PMID 17505218
- [Result] Bodey GP, Buckley M, Sathe YS, Freireich EJ. Quantitative relationships between circulating leukocytes and infection in patients with acute leukemia. Ann Intern Med. 1966 Feb;64(2):328-40. doi: 10.7326/0003-4819-64-2-328. No abstract available. PMID 5216294
- [Result] Lu M, Cao DM, Li DM, Zhao XX, Li JW, Li HX, Zhang HH, Zhang HF. [Effects of acupuncture and moxibustion on DNA excision repair-related proteins of bone marrow cell in cyclophosphamide-induced mice]. Zhongguo Zhen Jiu. 2009 Oct;29(10):821-4. Chinese. PMID 19873920
- [Result] Lu M, Cao DM, Zhao XX. [Study on dynamic effect of acupuncture on marrow cell cycle regulatory protein cyclin D1 expression and cell cycle in mice with cyclophosphamide induced myelosuppression]. Zhongguo Zhong Xi Yi Jie He Za Zhi. 2011 Feb;31(2):238-43. Chinese. PMID 21425582
- [Result] Lu W, Matulonis UA, Doherty-Gilman A, Lee H, Dean-Clower E, Rosulek A, Gibson C, Goodman A, Davis RB, Buring JE, Wayne PM, Rosenthal DS, Penson RT. Acupuncture for chemotherapy-induced neutropenia in patients with gynecologic malignancies: a pilot randomized, sham-controlled clinical trial. J Altern Complement Med. 2009 Jul;15(7):745-53. doi: 10.1089/acm.2008.0589. PMID 19552597
- [Result] Ye F, Liu D, Wang S, Xu L. Effects of electro-acupuncture on T cell subpopulations, NK activity, humoral immunity and leukocyte count in patients undergoing chemotherapy. J Tradit Chin Med. 2007 Mar;27(1):19-21. PMID 17393618
- [Result] Han YF, Gong Z, Huang LQ, Xia X, Zhao WJ. [Clinical study on acupuncture for leukopenia induced by chemotherapy]. Zhongguo Zhen Jiu. 2010 Oct;30(10):802-5. Chinese. PMID 21058473
- [Result] Yeh CH, Chien LC, Chiang YC, Lin SW, Huang CK, Ren D. Reduction in nausea and vomiting in children undergoing cancer chemotherapy by either appropriate or sham auricular acupuncture points with standard care. J Altern Complement Med. 2012 Apr;18(4):334-40. doi: 10.1089/acm.2011.0102. PMID 22515794